CLINICAL TRIAL: NCT00156546
Title: Evaluation of the Effectiveness of Antibiotic Prophylaxis in Children With a History of Upper Urinary Tract Infections:a Multicentre Randomised Study
Brief Title: Evaluation of the Effectiveness of Antibiotic Prophylaxis in Children With a Previous Urinary Tract Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Padova (Other)
Collaborators: Regione Veneto (Other); IL Sogno di Stefano (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRIS 2
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-09

CONDITIONS: Urinary Tract Infections
Keywords: Urinary tract infections; Children; Antibiotic prophylaxis; Renal scintigraphy; Vesico ureteral reflux
MeSH Terms: conditions — Urinary Tract Infections; Vesico-Ureteral Reflux

INTERVENTIONS:
Drug: antibiotic to reduce the recurrence of infection

SUMMARY:
Our hypothesis is that long-term antimicrobial prophylaxis does not reduce the recurrence of infection and the risk of appearance of kidney scars in children with a documented previous upper UTI.

DETAILED DESCRIPTION:
Background

Upper urinary tract infections (UTI) are common in children, especially when functional and anatomical abnormalities of the urinary tract co-exist, such as vesico-ureteral reflux (VUR), urinary tract obstruction uropathy and bladder dysfunction. They are associated with the risk of long-term complications, including permanent renal damage (renal scarring), which occurs in 15% of cases. The objective of the diagnosis and medical treatment of UTI in children is the prevention of such complications. Medical treatment includes long-term antimicrobial prophylaxis to be continued for periods ranging from 6 months to 2 years. Recent studies have revealed the emergence of therapy-induced resistance. A review of the literature has highlighted the lack of properly designed, large clinical trials, demonstrating the efficacy of long-term low-dose antimicrobial prophylaxis in terms of reduction in UTI recurrence.

Methods and design

The study is a controlled, randomised, open-label, 3-armed, parallel-group clinical trial comparing no prophylaxis (group 1) with prophylaxis with co-trimoxazole 15 mg/kg daily (group 2) and with amoxicillin + clavulanic acid 15 mg/kg daily (group 3) for 12 months.

Assuming that the incidence of recurrences is 20%, defining efficacy as an incidence of 10% per group and setting  error = 0.05 and power = 90%, 220 patients per group (i.e. a total of 660 patients) are required The study population will consist of children aged between 2 months and 6 years, with normal renal function (creatinine clearance  70 ml/min/1.73m2) and a first episode of documented UTI, who presents at least one of the following: an acute pyelonephritic lesion at the DMSA scan and/or a VUR at the baseline micturating cystography.

Patients will be followed-up for 12 months. Urinalysis and urine cultures will be performed every month and clinical examinations after 6 and 12 months; both will be performed whenever UTI is suspected. Sonography, Doppler sonography (optional) and DMSA scintigraphy will be performed at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 months and 6 years
* Creatinine clearance (calculated according to Schwartz)  70 ml/min/1.73 m2 (for children in their first year of life, serum creatinine levels within normal range for age and sex)
* First documented upper UTI (diagnostic criteria in Table 1)
* Imaging Diagnostic work-up completed (Table 2) with at least the presence of an acute lesion at the DMSA scan and or a primary non severe reflux ( 1st or 3rd degree)
* Informed consent of parents

Exclusion Criteria:

* Patients with chronic renal insufficiency or  30% relative function of one kidney at DMSA scan
* Patients with urinary tract disorders, such as vesico-ureteral reflux due to complex malformations of the urinary tract, obstruction of the posterior urethra, ureterocele or single kidney, neurogenic bladder
* Patients with reflux  4th degree
* Patients with pyelonephritis that developed during prophylaxis instituted because of prenatal diagnosis of urinary tract dilatation  Hypersensitivity to one of the two selected antimicrobial agents

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 660
Dates: Start 2000-05; Study Completion 2006-07

PRIMARY OUTCOMES:
The primary end-point is UTI Recurrence Rate during the 12-month observation period and the Development of renal damage (parenchymal scar) after 12 months.

SECONDARY OUTCOMES:
The secondary objectives are the comparison, in terms of efficacy and effectiveness, between two antimicrobial agents that are currently approved for prophylactic use: co-trimoxazole 15 mg/kg daily versus amoxicillin + clavulanic acid 15 mg/kg daily.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Zacchello, Professor, Study Chair — Departement of Pediatrics, University of Padova; Antonella Toffolo, Dr, Principal Investigator — Pediatric Unit Ospedale di Oderzo (TV) Italy; Alessandro Calderan, Dr, Principal Investigator; Giovanni Montini, Dr, Principal Investigator — Nephrology, Dialysis and Transplant Unit, Pediatric Departement, Azienda Ospedaliera-Università, Padova
Locations (16):
- Italy (16):
  - Pediatric Unit, Ospedale di Belluno, Belluno, Belluno
  - Pediatric Unit, Ospedale di Bentivoglio, Bentivoglio, Bologna
  - - Pediatric Department, Ospedale di Bolzano, Bolzano, Bolzano
  - Pediatric Unit, Ospedale di Cuneo, Cuneo, Cuneo
  - Pediatric Unit, Ospedale di Este - Monselice, Monselice, Padova
  - Nephrology, Dialysis and transplant Unit Pediatric Depatment,, Padua, Padova
  - Pediatric Unit, Ospedale di Piove di Sacco e Chioggia, Piove di Sacco, Padova
  - Pediatric Unit, Ospedale di Ravenna, Ravenna, Ravenna
  - Pediatric Unit, Ospedale di Castelfranco, Castelfranco Veneto, Treviso
  - Pediatric Unit, Ospedale di Motta di Livenza, Motta Di Livenza Oderzo, Treviso
  - Pediatric Unit, Ospedale di Dolo, Dolo, Venezia
  - Pediatric Unit, Ospedale di Soave, Soave, Verona
  - Pediatric Unit, Ospedale di Schio/Thiene, Thiene, Vicenza
  - Pediatric Department, Ospedale Maggiore, Bologna
  - Pediatric Unit, Ospedale di Mestre, Mestre Venezia
  - Pediatric Unit, Ospedale di Verona, Verona

REFERENCES:
- [Background] Chon CH, Lai FC, Shortliffe LM. Pediatric urinary tract infections. Pediatr Clin North Am. 2001 Dec;48(6):1441-59. doi: 10.1016/s0031-3955(05)70385-0. PMID 11732124
- [Background] Benfield MR, McDonald R, Sullivan EK, Stablein DM, Tejani A. The 1997 Annual Renal Transplantation in Children Report of the North American Pediatric Renal Transplant Cooperative Study (NAPRTCS). Pediatr Transplant. 1999 May;3(2):152-67. doi: 10.1034/j.1399-3046.1999.00011.x. PMID 10389139
- [Background] Wennerstrom M, Hansson S, Jodal U, Stokland E. Primary and acquired renal scarring in boys and girls with urinary tract infection. J Pediatr. 2000 Jan;136(1):30-4. doi: 10.1016/s0022-3476(00)90045-3. PMID 10636970
- [Background] Hoberman A, Wald ER, Hickey RW, Baskin M, Charron M, Majd M, Kearney DH, Reynolds EA, Ruley J, Janosky JE. Oral versus initial intravenous therapy for urinary tract infections in young febrile children. Pediatrics. 1999 Jul;104(1 Pt 1):79-86. doi: 10.1542/peds.104.1.79. PMID 10390264
- [Background] Downs SM. Technical report: urinary tract infections in febrile infants and young children. The Urinary Tract Subcommittee of the American Academy of Pediatrics Committee on Quality Improvement. Pediatrics. 1999 Apr;103(4):e54. doi: 10.1542/peds.103.4.e54. PMID 10103346
- [Background] Hohenfellner K, Hunley TE, Brezinska R, Brodhag P, Shyr Y, Brenner W, Habermehl P, Kon V. ACE I/D gene polymorphism predicts renal damage in congenital uropathies. Pediatr Nephrol. 1999 Aug;13(6):514-8. doi: 10.1007/s004670050649. PMID 10452281
- [Background] Bollgren I. Antibacterial prophylaxis in children with urinary tract infection. Acta Paediatr Suppl. 1999 Nov;88(431):48-52. doi: 10.1111/j.1651-2227.1999.tb01318.x. PMID 10588271
- [Background] Williams G, Lee A, Craig J. Antibiotics for the prevention of urinary tract infection in children: A systematic review of randomized controlled trials. J Pediatr. 2001 Jun;138(6):868-74. doi: 10.1067/mpd.2001.113785. PMID 11391331
- [Background] Williams GJ, Lee A, Craig JC. Long-term antibiotics for preventing recurrent urinary tract infection in children. Cochrane Database Syst Rev. 2001;(4):CD001534. doi: 10.1002/14651858.CD001534. PMID 11687116
- [Background] Ghiro L, Cracco AT, Sartor M, Comacchio S, Zacchello G, Dall'Amico R; Veneto Urinary Tract Infection Study Group. Retrospective study of children with acute pyelonephritis. Evaluation of bacterial etiology, antimicrobial susceptibility, drug management and imaging studies. Nephron. 2002 Jan;90(1):8-15. doi: 10.1159/000046308. PMID 11744799
- [Derived] Montini G, Rigon L, Zucchetta P, Fregonese F, Toffolo A, Gobber D, Cecchin D, Pavanello L, Molinari PP, Maschio F, Zanchetta S, Cassar W, Casadio L, Crivellaro C, Fortunati P, Corsini A, Calderan A, Comacchio S, Tommasi L, Hewitt IK, Da Dalt L, Zacchello G, Dall'Amico R; IRIS Group. Prophylaxis after first febrile urinary tract infection in children? A multicenter, randomized, controlled, noninferiority trial. Pediatrics. 2008 Nov;122(5):1064-71. doi: 10.1542/peds.2007-3770. PMID 18977988
- [Derived] Hewitt IK, Zucchetta P, Rigon L, Maschio F, Molinari PP, Tomasi L, Toffolo A, Pavanello L, Crivellaro C, Bellato S, Montini G. Early treatment of acute pyelonephritis in children fails to reduce renal scarring: data from the Italian Renal Infection Study Trials. Pediatrics. 2008 Sep;122(3):486-90. doi: 10.1542/peds.2007-2894. PMID 18762516